CLINICAL TRIAL: NCT06068309
Title: Perception, Adherence, Clinical, Economical and Health-Related Quality of Life Outcomes of CareAide® App Usage in Chronic Diseases
Brief Title: Efficacy of CareAide® App in Improving Adherence in Adults With Chronic Diseases
Acronym: CAREAide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Caring Up Pte Ltd, Malaysia (Unknown); Institute of Adherence to Medication, American University of Health Sciences, United States (Unknown)
Responsible Party: Principal Investigator, Dr. Rajat Rana, Clinical Trial Researcher, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMRR ID-22-01108-COI; UM.0000532/HPV.PV (Other Grant/Funding Number: Caring Up Malaysia Pte. Ltd., 50470 Kuala Lumpur. Malaysia)
Record Dates: First submitted 2023-09-19; First posted 2023-10-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Adherence, Medication; Chronic Disease; Quality of Life; Economic Burden; Asthma; Hypertension; Heart Failure; Diabetes
Keywords: randomized controlled trial; mobile health app; digital health; medication adherence app; Patient perception; CareAide; clinical outcomes; Malaysia; adherence
MeSH Terms: conditions — Medication Adherence; Chronic Disease; Financial Stress; Asthma; Hypertension; Heart Failure; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CareAide Interventional Group (Experimental): Participants allocated to the Interventional group (IG) uses the CareAide® app on their smartphones in addition to prescribed usual therapeutic care.
  Interventions: Other: CareAide App Usage
- Control Group (No Intervention): Participants allocated to the Control group (CG) receives prescibed usual therapeutic care

INTERVENTIONS:
Other: CareAide App Usage — The study participant uses the CareAide app in addition to prescribed usual therapeutic care
  Arms: CareAide Interventional Group

SUMMARY:
The goal of this clinical trial is to study the impact of a medication adherence app, CareAide, in adult population diagnosed with chronic diseases in Malaysian population.

The main question[s] it aims to answer are:

1. Can CareAide make people take their medications better and improve their health?
2. Can CareAide improve the health of people with chronic diseases?
3. Does using CareAide make people's lives better?
4. Can CareAide save money when managing chronic diseases?
5. How do people feel about using CareAide?

Researchers will ask the participants to use the CareAide app for 6 months and compare the group that used the app with the other group which just received the usual treatment. Researchers will check if they do better with their medications, feel healthier, have a better life, and spend less money. They will check this twice, once after 3 months and again after 6 months.

adherence, clinical outcomes, quality of life and economic associated with the app with two follow ups at 3 month intervals.

DETAILED DESCRIPTION:
According to WHO and Ministry of Health (MOH) Malaysia 2020 report, expenditure for chronic diseasesestimated involved around 0.65% of Malaysia's gross domestic product (GDP) which is about RM8.91 billion (Ministry of Health Malaysia, 2020). This showed that chronic diseases imposed a significant healthburden to our country. Malaysian population having good and easy access to effective medical therapyunder the public healthcare system, approximately 46% to 56% of patients with hypertension were non-adherent in terms of their medications. Therefore, CareAide App will be used to study and identify the effect, clinical outcome and cost effectiveness of mobile health app in managing chronic diseases.

The Comprehensive Adherence-enhancing Reminder and Engagement Aide (CAREAide) Trial aims to assess the effect of CareAide® app on adherence, clinical outcomes of patients with chronic diseases and user's perception and satisfaction with the app.

A 3-and 6- month open-label multicentre randomized controlled trial with two parallel groups will be conducted. This study will take place in the outpatient setting of the three hospitals [i.e., Hospital Putrajaya, Hospital Pulau Pinang and Universiti Malaya Medical Center (UMMC)) in Malaysia]. Both interventional and control group will be allocated to 1:1 ratio. Randomization number will be generated by using online number generated programme. Consultants reviewing patients at medical, cardiology,diabetes mellitus and asthma clinics will provide referral and notify independent researchers for eligibility and group assignments. Eligible patients will then be instructed to see pharmacists/researchers atoutpatient pharmacies to refill their prescriptions and subsequently enrol in the assigned study group either to receive an intervention with CareAide® or to receive normal clinical care. Information and training on the app will be provided by these researchers to the participants.Patients will be recruited at therespective outpatient clinics. At the usual care clinic appointments, patients have their demographics and baseline data of blood pressure, blood sugar, basic blood profiles, asthma control and review of theirdisease management collected by consultants/researchers. Patients who meet the study criteria will then be instructed to see pharmacists/researchers at outpatient pharmacy to refill their medications. The pharmacists/researchers will screen patients' inclusion and exclusion criteria for this study and will explainthat they may or may not be selected for the study and if they agree, proceed to provide written informedconsent. The adherence data from the screening will be collected to gauge the general adherence rate inthese group of patients. An independent researcher, who is not involved in the intervention and controlgroups, will use the random number generator software for randomisation sequences. The random numbers will be placed in opaque envelopes, which subsequently will be opened by pharmacists/researchers at the outpatient pharmacies. Participants and pharmacists/researchers are unblinded to group assignment and are aware of the intervention, but the study hypotheses are not disclosed to the participants. The assessor and statisticians are blinded to participant allocation. The study will be evaluating usual care compared with usual care plus pharmacist-driven patient-specific adherence interventions - CareAide® medication adherence digital application. Usual care provided bythese hospitals comprises clinic appointments every 3 to 6 months. Medication adherence: CareAide® effectiveness is measured with a medication adherence tool at baseline and follow-up time periods at 3months and 6 months using Morisky Medication Adherence Scale (MMAS) and proportion of days covered (PDC). MMAS-8 is a licensed validated questionnaire to assess medication adherence, where a higher score represents higher medication adherence and vice versa. Comprising of 8 items, the score ranges from 0 to 8, where a higher score represents a higher medication adherence. The internal consistency (Cronbach's alpha) of MMAS-8 is 0.83 along with a sensitivity of 93% and a specificity of 57%.

The PDC method utilises pharmacy refill records. Fasting blood sugar, HbA1C, cardiovascular events (heart failure admission, mortality), asthma control and blood pressure, hospitalizations and emergency visits measurements will be based on the clinics attended by the participants. Health care utilization, quality of life and health care expenditures willbe measured for all the participants.

Intention to treat (ITT) analysis will be applied to evaluate the results to avoid any bias. The data analysiswill be using the SPSS version 29. Data will be coded and analysed. Descriptive or categorical data will beexpressed as mean ± standard deviation (SD) unless otherwise stated. Student t-test will be used foranalysis of normally distributed or continuous variables. Mann-Whitney test will be used for non-normallydistributed data. Categorical data will be analysed using Chi-square or Fischer's exact test. A value of P <0.05 is considered statistically significant.

The prevalence of medication compliant is quantified at 3 months and 6 months follow-up. Independent t-test or Mann-Whitney test will be used to compare MMAS score rankings between the intervention andcontrol groups. Chi-Square test of independence will be used to determine the difference in number ofpatients with medication adherence between the intervention and control groups at 3 months and 6months follow-up. Ordinal logistic regression, with the MMAS adherence score ranking, will be used to examine the association between intervention and control groups.

For the perception and satisfaction towards the app, the frequency and percentage of respondents in each category (strongly disagree to strongly agree) will be calculated. The median of each statement will then be calculated to give an overview of perception and satisfaction towards the CareAide® app. Chi-square, Mann-Whitney U, Kriskall Wallis, Chi-square tests and logistic regression will be used where appropriate. Linear regression analysis will be conducted to determine the independent predictors of HRQoL.

An economic evaluation will be conducted from a payer and societal perspective. Costs and outcomes will be discounted at 3% per year as the results will be extrapolated to examine costs and outcome over a year. Cost effectiveness analysis will be estimated based on the results of cost data and the incremental cost per quality adjusted life year (QALY) gained. Total incremental cost effectiveness ratio (ICER) will be calculated by dividing the difference between the cost of CareAide intervention group and control group by the difference between the QALYs of CareAide intervention group and control group. Sensitivity analysis will be performed by bootstrapping technique to ensure or examine the robustness of ICER. Then, cost effectiveness acceptability curve (CEAC) will be created to estimate the proportion of the result being cost-effective in relation to the Willingness-to-Pay (WTP) threshold.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and above
* Diagnosed with selected non-communicable diseases (NCDs): hypertension, diabetes mellitus, heart failure or asthma for at least 6 months
* Prescription generated from one of the following specialty clinics: Medical, Cardiology, Diabetes Mellitus or Asthma clinics of study site.
* Medications are prescribed in previous 3 months and refill at the point of recruitment
* Morisky Medication Adherence Scale (MMAS) score < 6 (i.e. Low adherence)
* More than three medications daily or two medications with multiple dosing intervals.
* One or more hospital admissions in the prior 24 months
* Owns a smartphone

Exclusion Criteria:

* Medications prescribed from other institution providers
* Existing mobile health app or medication reminder app user
* Pregnant
* Cognitively impaired
* Prisoners
* Bed-bound
* Severe diseases/comorbidities - terminal cancer, psychiatry, etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2022-07-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Morisky Medication Adherence Scale (MMAS) Score | 6 Months
  Adherence measured by the 8-item Morisky Medication Adherence Scale (MMAS-8) where a scoring is as defined as, Low Adherence (0< 6); Medium Adherence (6 to <8); High Adherence (= 8)
Proportion of days covered (PDC) | 6 Months
  Adherence is measured by Proportion of days covered (PDC) which measures the proportion of days in which a subject has access to their medication over a specified period of time (POI). It is calculated as the (sum of days covered in the POI) ÷ (number of days in the POI) × 100, Scoring is defined as, High adherence (>80%); Medium Adherence (50%-80%); Poor adherence (<50%)

SECONDARY OUTCOMES:
Clinical Parameter of Hypertension: Blood Pressure | 6 Months
  Hypertensive clinical parameters, Systolic blood pressure (SBP) and Diastolic blood pressure (DBP) are measured, where SBP (≥140 mm Hg); DBP (≥90 mm Hg) levels are considered Hypertensive.
Clinical Parameter of Heart Failure: Ejection fraction | 6 Months
  Ejection fraction (EF) is a measurement, expressed as a percentage, of how much blood the left ventricle pumps out with each contraction. It is classified as Reduced (EF≤40%); Borderline (EF≈41-49%); Normal (EF≈50-70%).
Clinical Parameter of Diabetes: Glycated hemoglobin | 6 Months
  Glycated hemoglobin (HbA1c) is measured for diagnosis of Diabetes, where a patient with HbA1c >6.5% is considered Diabetic.
Clinical Parameter of Diabetes: Glucose levels | 6 Months
  Glucose levels, specifically Fasting blood glucose (FBG) (>125 mg/dL), Random blood glucose (RBG) (>200 mg/dL) and Post-Prandial blood glucose PPBG at 2 hours (>200 mg/dl) are indicative of diabetic.
Clinical Parameter of Asthma: Forced Expiratory Volume in 1 second | 6 Months
  Forced expiratory volume in 1 second (FEV1) is the maximum amount of air that the subject can forcibly expel during the first second following maximal inhalation. A patient is considered a high risk if FEV1 is less than 60% and Low risk if his FEV1 is more than 60%.
Clinical Parameter of Asthma: Peak Expiratory Flow | 6 Months
  Peak expiratory flow (PEF) is the maximum flow rate (expressed in liters per minute [L/min]) generated during a forceful exhalation, starting from full inspiration. It is classified as Persistent Asthma with symptoms (Severe Persistent (PEF<60%); Moderate Persistent (PEF 60-79%); Mild Persistent (PEF>80%), Intermittent Asthma without symptoms (PEF>80%))
Clinical Parameter of Asthma: Asthma Control Questionnaire-7 (ACQ-7) Score | 6 Months
  The ACQ score ranges between 0 (well controlled) and 6 (extremely poorly controlled). It classifies asthma control as well controlled (≤0.75); Inadequately controlled (≥1.5); Minimal important difference (0.5).
Total Medical Cost | 6 Months
  Total Medical Cost will be calculated in Malaysia currency, Ringgit Malaysia (RM). It will involve direct, indirect, and intangible costs. Direct cost refers to the costs incurred because of medical management of the disease, drugs, admissions, complementary tests, patient transportation. The Indirect costs refers to the costs incurred not as a result of medical management of the disease but rather of other incurred losses such as lost wages, lost productivity, and costs resulting from the need for home care and child care that would otherwise not be incurred. Intangible costs are those associated with the function lost, increased pain and reduced life quality.
Incremental Cost-Effectiveness Ratio (ICER) | 6 Months
  The ICER is calculated as the difference in the expected costs of the two health interventions i.e. CareAide app users with usual therapeutic care versus only usual therapeutic standard care, divided by the difference in their expected effects i.e. improvement in adherence (QALYs).
Health-related quality of life (HRQoL): EuroQol-5D (EQ-5D-5L) Questionnaire | 6 Months
  The EQ-5D-5L comprises two pages: the descriptive system (five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; each with five levels) and the EQ VAS (a vertical scale indicating self-rated health from 'best health imaginable' to 'worst health imaginable'). The patient marks their health state by choosing a statement for each dimension, resulting in a 5-digit number. The EQ VAS serves as a quantitative measure of the patient's health judgment..
Health-related quality of life (HRQoL): Short-form (SF-36) Survey Instrument | 6 Months
  A 36-item short-form (SF-36) was constructed to survey health status in the Medical Outcomes Study. The self-administered SF-36 includes one multi-item scale that assesses eight health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions.
Perception & Satisfaction Questionnaire (PSQ) | 6 Months
  Only the participants using the CareAide® app will be given Perception & Satisfaction Questionnaire (PSQ) at the end of 6 months follow up to understand the participant's perception of the perceived usefulness of the app and rate their satisfaction with the app. The questionnaire will be divided into three sections to specify the type of questions to be asked. The first section consists of basic demographics, including age, gender, ethnicity, personal health status, and the number of medications taken. Section two includes questions to explore the perception of the users towards the app. Section three consists of a questionnaire to rate their satisfaction with the app. The responses will be measured using a 5-point Likert scale with score ranging from 1 (Inadequate) to 5 (Excellent)

CONTACTS AND LOCATIONS:
Overall Officials: Ong Siew Chin, PhD, Principal Investigator — School of Pharmaceutical Sciences, Universiti Sains Malaysia (USM), Penang, Malaysia; Navin Kumar Loganadan, PhD, Principal Investigator — Hospital Putrajaya, Malaysia; Jaya Muneswarao M Devudu, Principal Investigator — Hospital Pulau Pinang, Malaysia; Izyan A Wahab, PhD, Principal Investigator — Faculty of Pharmacy, University of Malaya, 50603 Kuala Lumpur, Malaysia; Kayatri Govindaraju, PhD, Principal Investigator — Faculty of Pharmacy, University of Malaya, 50603 Kuala Lumpur, Malaysia; Rajat Rana, Pharm.D, Principal Investigator — Faculty of Pharmacy, University of Malaya, 50603 Kuala Lumpur, Malaysia; Ng Chow Kyn, MPharm Clin, Principal Investigator — School of Pharmaceutical Sciences, Universiti Sains Malaysia (USM), Penang, Malaysia; Mohamed Syamir Shukeri, MCH, Principal Investigator — Faculty of Pharmacy, University of Malaya, 50603 Kuala Lumpur, Malaysia; Baharudin Ibrahim, PhD, Principal Investigator — Faculty of Pharmacy, University of Malaya, 50603 Kuala Lumpur, Malaysia; Hasniza Zaman Huri, PhD, Principal Investigator — Faculty of Pharmacy, University of Malaya, 50603 Kuala Lumpur, Malaysia
Locations (3):
- Malaysia (3):
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Putrajaya, Putrajaya

REFERENCES:
- [Background] Asche C, LaFleur J, Conner C. A review of diabetes treatment adherence and the association with clinical and economic outcomes. Clin Ther. 2011 Jan;33(1):74-109. doi: 10.1016/j.clinthera.2011.01.019. PMID 21397776
- [Background] Baker-Eveleth, L., & Stone, R. W. (2020). User's perceptions of perceived usefulness, satisfaction, and intentions of mobile application. International Journal of Mobile Communications, 18(1), 1-18.
- [Background] Charan J, Biswas T. How to calculate sample size for different study designs in medical research? Indian J Psychol Med. 2013 Apr;35(2):121-6. doi: 10.4103/0253-7176.116232. PMID 24049221
- [Background] Cano Martin JA, Martinez-Perez B, de la Torre-Diez I, Lopez-Coronado M. Economic impact assessment from the use of a mobile app for the self-management of heart diseases by patients with heart failure in a Spanish region. J Med Syst. 2014 Sep;38(9):96. doi: 10.1007/s10916-014-0096-z. Epub 2014 Jul 4. PMID 24994514
- [Background] Chia YC, Devaraj NK, Ching SM, Ooi PB, Chew MT, Chew BN, Mohamed M, Lim HM, Beh HC, Othman AS, Husin HS, Mohamad Gani AH, Hamid D, Kang PS, Tay CL, Wong PF, Hassan H. Relationship of an adherence score with blood pressure control status among patients with hypertension and their determinants: Findings from a nationwide blood pressure screening program. J Clin Hypertens (Greenwich). 2021 Mar;23(3):638-645. doi: 10.1111/jch.14212. Epub 2021 Feb 14. PMID 33586334
- [Background] Consort - The CONSORT Flow Diagram. (2021). Retrieved 11 December 2021, from http://www.consort-statement.org/consort-statement/flow-diagram.
- [Background] Eysenbach G; CONSORT-EHEALTH Group. CONSORT-EHEALTH: improving and standardizing evaluation reports of Web-based and mobile health interventions. J Med Internet Res. 2011 Dec 31;13(4):e126. doi: 10.2196/jmir.1923. PMID 22209829
- [Background] Islam, S., Peiffer, R., Chow, C., Maddison, R., Lechner, A., & Holle, R. et al. (2020). Cost-effectiveness of a mobile-phone text messaging intervention on type 2 diabetes-A randomized-controlled trial. Health Policy and Technology, 9(1), 79-85
- [Background] Vahatalo I, Kankaanranta H, Tuomisto LE, Niemela O, Lehtimaki L, Ilmarinen P. Long-term adherence to inhaled corticosteroids and asthma control in adult-onset asthma. ERJ Open Res. 2021 Feb 8;7(1):00715-2020. doi: 10.1183/23120541.00715-2020. eCollection 2021 Jan. PMID 33585657
- [Background] Li J, Sun L, Hou Y, Chen L. Cost-Effectiveness Analysis of a Mobile-Based Intervention for Patients with Type 2 Diabetes Mellitus. Int J Endocrinol. 2021 Jul 1;2021:8827629. doi: 10.1155/2021/8827629. eCollection 2021. PMID 34306072
- [Background] Lins L, Carvalho FM. SF-36 total score as a single measure of health-related quality of life: Scoping review. SAGE Open Med. 2016 Oct 4;4:2050312116671725. doi: 10.1177/2050312116671725. eCollection 2016. PMID 27757230
- [Background] Melin J, Bonn SE, Pendrill L, Trolle Lagerros Y. A Questionnaire for Assessing User Satisfaction With Mobile Health Apps: Development Using Rasch Measurement Theory. JMIR Mhealth Uhealth. 2020 May 26;8(5):e15909. doi: 10.2196/15909. PMID 32452817
- [Background] Perez-Jover V, Sala-Gonzalez M, Guilabert M, Mira JJ. Mobile Apps for Increasing Treatment Adherence: Systematic Review. J Med Internet Res. 2019 Jun 18;21(6):e12505. doi: 10.2196/12505. PMID 31215517
- [Background] Purcell R, McInnes S, Halcomb EJ. Telemonitoring can assist in managing cardiovascular disease in primary care: a systematic review of systematic reviews. BMC Fam Pract. 2014 Mar 7;15:43. doi: 10.1186/1471-2296-15-43. PMID 24606887
- [Background] Shang P, Liu GG, Zheng X, Ho PM, Hu S, Li J, Jiang Z, Li X, Bai X, Gao Y, Xing C, Wang Y, Normand SL, Krumholz HM. Association Between Medication Adherence and 1-Year Major Cardiovascular Adverse Events After Acute Myocardial Infarction in China. J Am Heart Assoc. 2019 May 7;8(9):e011793. doi: 10.1161/JAHA.118.011793. PMID 31057004
- [Background] Tsuji S, Ishikawa T, Morii Y, Zhang H, Suzuki T, Tanikawa T, Nakaya J, Ogasawara K. Cost-Effectiveness of a Continuous Glucose Monitoring Mobile App for Patients With Type 2 Diabetes Mellitus: Analysis Simulation. J Med Internet Res. 2020 Sep 17;22(9):e16053. doi: 10.2196/16053. PMID 32940613
- [Background] Wood AM, White IR, Thompson SG. Are missing outcome data adequately handled? A review of published randomized controlled trials in major medical journals. Clin Trials. 2004;1(4):368-76. doi: 10.1191/1740774504cn032oa. PMID 16279275
- [Background] Juniper EF, Bousquet J, Abetz L, Bateman ED; GOAL Committee. Identifying 'well-controlled' and 'not well-controlled' asthma using the Asthma Control Questionnaire. Respir Med. 2006 Apr;100(4):616-21. doi: 10.1016/j.rmed.2005.08.012. Epub 2005 Oct 13. PMID 16226443
- [Background] Nau DP. Proportion of days covered (PDC) as a preferred method of measuring medication adherence. Springfield, VA: Pharmacy Quality Alliance. 2012;6:25.
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Background] Morisky DE, DiMatteo MR. Improving the measurement of self-reported medication nonadherence: response to authors. J Clin Epidemiol. 2011 Mar;64(3):255-7; discussion 258-63. doi: 10.1016/j.jclinepi.2010.09.002. Epub 2010 Dec 8. No abstract available. PMID 21144706

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-07-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT06068309/Prot_SAP_ICF_000.pdf